CLINICAL TRIAL: NCT04855188
Title: A Randomized, Multicenter, Evaluator-Blinded, Active-Controlled, Parallel-Group Design Investigation to Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 540 Versus YVOIRE Volume Plus in Nasolabial Folds Injection
Brief Title: Effectiveness and Safety of YVOIRE Y-Solution 540
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LG-HACL027
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Wrinkles in the Nasolabial Folds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YVOIRE Y-Solution 540 (Experimental)
  Interventions: Device: YVOIRE Y-Solution 540
- YVOIRE volume plus (Active Comparator)
  Interventions: Device: YVOIRE volume plus

INTERVENTIONS:
Device: YVOIRE Y-Solution 540 — Injection into the deep dermis layer and/or subcutaneous layer in the nasolabial folds based on the randomization assignment.
  Arms: YVOIRE Y-Solution 540
Device: YVOIRE volume plus — Injection into the deep dermis layer and/or subcutaneous layer in the nasolabial folds based on the randomization assignment.
  Arms: YVOIRE volume plus

SUMMARY:
To Evaluate the Effectiveness and Safety of YVOIRE Y-Solution 540 versus YVOIRE volume plus in Nasolabial Folds Injection

ELIGIBILITY:
Inclusion Criteria:

* 3 (moderate) or 4 (severe) on the 5-graded WSRS
* who sign the written informed consent form

Exclusion Criteria:

* who have received permanent facial implants
* who have received semi-permanent fillers
* who have undergone temporary dermal filler treatment within 12 months
* who have undergone facial tissue augmentation with fat injections, botulinum toxin injections, mesotherapy, or cosmetic procedures within 6 months
* who have a history of anaphylaxis or allergy to lidocaine, hyaluronic acid (HA) products, or streptococcal protein

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
WSRS responder rate | 24 weeks after the last injection
  the proportion of subjects with ≥ 1 grade improvement on the wrinkle severity rating scale (WSRS) score

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China